CLINICAL TRIAL: NCT05569980
Title: The Nordic Rectal Prolapse Study - a Multicentre, International Cohort Study
Brief Title: The Nordic Rectal Prolapse Study
Acronym: NORDIC
Status: Enrolling by invitation | Type: Observational
Sponsor: Aarhus University Hospital (Other)
Collaborators: Novo Nordisk A/S (Industry); Esbjerg Hospital - University Hospital of Southern Denmark (Other); Universitätsmedizin Mannheim (Other); Odense University Hospital (Other); Hillerod Hospital, Denmark (Other); Groene Hart Ziekenhuis (Other); ASZ Aalst (Other)
Responsible Party: Principal Investigator, Andreea-Alexandra Bach-Nielsen, Ph.D. student, Aarhus University Hospital
Other Study IDs: NORDIC
Record Dates: First submitted 2022-10-04; First posted 2022-10-06 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Rectal Prolapse; Surgery; Recurrence; Quality of Life
Keywords: Surgery; Recurrence; Quality of life; Bowel function
MeSH Terms: conditions — Rectal Prolapse; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to gather data about surgical procedures for rectal prolapse in adult human subjects. The main question it aims to answer is:

• Which procedure is best for treating external rectal prolapse?

Participants will:

* be included if they can consent to participation
* be offered standard care treatment, as no interventions will be done
* be asked to answer relevant questionnaires within 3 months prior to the surgery for rectal prolapse
* be asked to answer the same questionnaires 6 and 12 months postoperative
* optionally answer the questionnaires again at 3 and 1 year postoperative, but this is not part of the existing funding body

DETAILED DESCRIPTION:
The Nordic Rectal Prolapse Study (NORDIC) is an observational trial initiated from the Pelvic Floor Unit, Aarhus University Hospital (AUH), planned in collaboration with the Pelvic Floor Society, UK. Although an RCT is the most favourable design for interventional surgical trials, it took seven years to recruit 75 patients for an RCT from Aarhus. Observational studies generally recruit with greater ease than RCTs, and this type of design is a valid option to an RCT. The non-randomized design can encourage inclusion as the type of surgery will be as per routine care, and the study is able to adapt to variations in practice during the trial period.

The investigators hypothesize that laparoscopic ventral mesh rectopexy (LVMR) is superior to other surgical procedures for rectal prolapse when it comes to improvement in quality of life for the patients.

Lead site will be the Department of Surgery, AUH. Expression of interest (EoI) forms have been collected from sites in Denmark, Scandinavia, and the UK. Patients undergoing rectal prolapse surgery will be eligible for inclusion respecting a few exclusion criteria. The trial is observational only. Surgical procedure will be by choice of the individual surgeon in collaboration with the patient. Thus, standard practice will be observed at different sites. Due to the high number of participating patients and surgical units, sufficient variation in procedures is assumed.

Quality of life measured by means of EQ-5D (European Quality of Life - 5 Dimensions) at 6 months postoperative will be the primary endpoint. There has been assumed 90% power to demonstrate non-inferiority with a two-sided 95% confidence interval, a non-inferiority margin of 0.1, a standard deviation of 0.26 based on UK population data, and that the correlation between baseline and follow-up EQ-5D is 0.4. Allowing for 10% loss to follow-up the researchers aim to recruit 430 participants in total. A conservative estimate assumes 20 centres with >15 eligible patients per year. With a recruitment rate of 80% the investigators should be able to recruit >480 patients over a 24-months period, allowing for staggered site initiation.

Data will be collected preoperative both from patient records and by patient reported outcome measures (PROMs) covering QoL, bowel function, urinary and sexual function, pain, and global satisfaction, and will be distributed electronically or on paper according to patient preferences.

Main assessment will be PROMs at defined time points.

ELIGIBILITY:
Inclusion Criteria:

• undergoing surgery for rectal prolapse

Exclusion Criteria:

• unable to consent to participating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients getting surgery for external rectal prolapse.
Sampling Method: Non-Probability Sample
Enrollment: 430 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Quality of life after surgery | 6 months
  To determine whether well-established procedures for external rectal prolapse are non-inferior to LVMR using EQ-5D at 6 months post-surgery.

SECONDARY OUTCOMES:
Constipation | 12 months
  To determine the effect of different procedures on constipation symptoms using PAC-SYM score at 6- and 12-months post-operatively.
Faecal incontinence | 6 months
  To determine the effect of different procedures on faecal incontinence (Wexner Score), MyMOP 2, and on single questions on urinary and sexual function, pain, global satisfaction at 6m.
Complications | 6 months
  To determine rates of short-term harms based on perioperative complications and medium-term follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Christensen, Prof., MDSc, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: No